CLINICAL TRIAL: NCT00512265
Title: Influence of N-Acetylcysteine on Morbidity, Oxygenation and Cytokine Levels in Partial or Total Esophagectomy for Cancer. A Multicenter, Prospective, Randomised Double Blind, Placebo-controlled Study
Brief Title: Influence of N-Acetylcysteine on Morbidity, Oxygenation and Cytokine Levels in Partial or Total Esophagectomy for Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Triemli Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005DR4333
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Pulmonary Morbidity
Keywords: n-acetylcysteine; esophagectomy; inflammatory reaction; pulmonary morbidity
MeSH Terms: conditions — Inflammation | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 150mg/kg N-Acetylcysteine in 250mL Glucose 5% at time of induction of anaesthesia 50mg/kg N-Acetylcysteine in 250mL Glucose 5% on post-op days 1-3
  Interventions: Drug: n-acetylcysteine
- 2 (Placebo Comparator): placebo (250mL glucose 5%) at time of induction of anaesthesia placebo (250mL glucose 5%) on post-op days 1-3
  Interventions: Drug: 250mL glucose 5%

INTERVENTIONS:
Drug: n-acetylcysteine — 150mg/kg N-Acetylcysteine in 250mL Glucose 5% at time of induction of anaesthesia 50mg/kg N-Acetylcysteine in 250mL Glucose 5% on post-op days 1-3
  Arms: 1
Drug: 250mL glucose 5% — placebo (250mL glucose 5%) at time of induction of anaesthesia placebo (250mL glucose 5%) on post-op days 1-3
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effect of high-dose n-acetylcysteine on inflammatory reaction, pulmonary morbidity, oxygenation and quality of life in patients undergoing transthoracic, partial or total resection of the esophagus for cancer.

DETAILED DESCRIPTION:
Cancer of the esophagus has a poor long term prognosis as well as high perioperative morbidity. Pulmonary complications play thereby a major role. The standard procedure is either a combined transabdominal/transthoracic approach, which allows better visualisation of the tumor and more radical surgery (which may increase R0 resections and consequently overall survival) or a blunt transhiatal technique. In Zurich, Basel and Lucerne, the combined technique is the standard procedure. The combined surgical approach, pre-existing pulmonary disorders, poor nutritional status and the release of pro-inflammatory cytokines may be important contributing factors to pulmonary complications such as pneumonia, atelectasis, pleural effusions and the Acute Respiratory Distress Syndrome (ARDS). N-Acetylcysteine (NAC) has been shown to have direct and indirect oxygen scavenging abilities. In severe sepsis and acute respiratory distress syndrome, positive effects of NAC on morbidity and mortality were discovered. Aim of this study is to assess the influence of NAC on morbidity, oxygenation parameters and cytokine levels.

According to power analysis, 90 patients have to be included in the trial. A multicenter approach was chosen to finish the study within 3 years. Respective to the average number of operations per institution and year, the following distribution is planned: Triemli Hospital 40, University Hospital Basel 30, Kantonsspital Lucerne 20. Inclusion criteria for this trial are patients undergoing thoraco-abdomino-cervical or abdomino-thoracic esophagectomy for cancer between 20 and 90 years and given informed consent. Exclusion criteria are known allergy or hypersensitivity to NAC and pregnancy. Patients are randomised to receive either high dose N-Acetylcysteine administered perioperatively and postoperatively for three days (150mg/kg perioperatively and 50mg/kg days 1-3) or placebo (glucose 5%).

Pre-, peri- and postoperatively cytokines (IL-1, IL-1ra, IL-6, IL-8, IL-10, TNF-α), are quantified by enzyme-linked immuno assay (ELISA) from blood, broncho-alveolar lavage and lavage of pleural space. Leucocytes, C-reactive protein, Procalcitonin and oxygenation parameters (arterial blood gas analyses = ABGA) are regularly measured. Morbidity and mortality is assessed. Furthermore, all patients are asked to complete a quality of life questionnaire (EORTC QLQ-OES18 and 30, SF-36) before and after the operation (12, 24, 36 months post-op).

ELIGIBILITY:
Inclusion Criteria:

* elective, abdomino-thoracic esophagectomy
* elective, thoraco-abdomino-cervical esophagectomy
* age 20-90 years
* informed consent given

Exclusion Criteria:

* emergency procedures
* patients with increased bronchorrhoea
* hypersensitivity against n-acetylcysteine
* pregnancy
* lactation

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Influence of n-acetylcysteine on inflammatory reaction measured by 1. cytokines in blood, broncho-alveolar lavage and pleural lavage; 2. postoperative course of Leucocytes, C - reactive protein and Procalcitonin. | 1 year

SECONDARY OUTCOMES:
Influence of NAC on peri- and postoperative oxygenation parameters pO2, pO2/FiO2 oxygenation index), pCO2, HCO3-, Base Excess, pH. | 1 year
Influence of NAC on postoperative morbidity and mortality. | 1 year
Long term analysis of quality of life after esophagectomy. | 5 years
Influence of NAC on peri- and postoperative oxygenation parameters pO2, pO2/FiO2 (oxygenation index), pCO2, HCO3-, Base Excess, pH. | 1 year
Compare inflammatory reaction left vs right lung and other compartments | 2 years from launch

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, PD, MD, Principal Investigator — University Hospital Basel, Switzerland, Dep. Surgery; Andreas Zollinger, MD, Study Director — Departement of Anaesthesia and Intensive Care,Triemli Hospital, Zurich, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Department of Surgery, Triemli Hospital, Zurich, Switzerland, Zurich